CLINICAL TRIAL: NCT00310791
Title: Effects of Adrenal and Gonadal Hormone Replacement in Young Women With Anorexia Nervosa
Brief Title: Adrenal and Gonadal Hormone Replacement in Anorexia Nervosa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine M. Gordon, Catherine Gordon, MD, MSc, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anorexia04; R01HD043869 (NIH); NCT01343771 (obsolete NCT alias)
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; adolescents; dual-energy x-ray absorptiometry; dehydroepiandrosterone (DHEA); osteoporosis
MeSH Terms: conditions — Anorexia Nervosa; Osteoporosis | interventions — Hormone Replacement Therapy; Estrogens; Progestins; Ethinyl Estradiol-Norgestrel Combination; Ethinyl Estradiol; Levonorgestrel; Estrogens, Conjugated (USP); Sugars; Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo (sugar pill); identical to treatment medication capsule
  Interventions: Other: Placebo (Sugar Pill)
- DHEA + Hormone replacement therapy (estrogen/progestin) (Experimental): Combined therapy of dehydroepiandrosterone (DHEA) and hormone replacement therapy (ERT). Patients randomized to the DHEA + HRT arm will receive micronized oral DHEA in a dose of 50 mg daily + HRT (0.3 mg Premarin, 1 tablet daily for 3 months, follow by Alesse (20 mg ethinyl estradiol + 0.1 mg levonorgestrel for 15 months). The estrogen/progestin component of the regimen has been chosen to maximize patient compliance, as patients with AN may experience bloating or nausea if higher estrogen doses (> 20 g) are initiated too rapidly. The DHEA capsule strength will be 50 mg, the total daily dose to be studied in combination with HRT. The micronized DHEA preparation achieves more constant DHEA and DHEA-S levels. Fifty milligrams appears to be a physiological replacement dose for these young women, determined both from our pilot (10) and longitudinal studies (7).
  Interventions: Drug: Hormone replacement therapy (estrogen/progestin); Drug: Dehydroepiandrosterone (DHEA)

INTERVENTIONS:
Drug: Hormone replacement therapy (estrogen/progestin) — Hormone replacement therapy (estrogen/progestin). 0.3 mg conjugated estrogens x 3 months, followed by 9 months of oral contraceptive (20 mg ethinyl estradiol + 0.1 mg levonorgestrel)
  Other Names: Alesse (20 mg ethinyl estradiol + 0.1 mg levonorgestrel); Premarin (conjugated estrogens)
  Arms: DHEA + Hormone replacement therapy (estrogen/progestin)
Other: Placebo (Sugar Pill) — Placebo (sugar pill)
  Other Names: Placebo; Sugar pill
  Arms: Sugar Pill
Drug: Dehydroepiandrosterone (DHEA) — 50 mg tablet, 1 daily
  Other Names: Prasterone
  Arms: DHEA + Hormone replacement therapy (estrogen/progestin)

SUMMARY:
This study seeks to gain new information on why young women with anorexia nervosa are predisposed to early bone loss and osteoporosis. Through a randomized treatment trial in which participants will receive either combined therapy with the adrenal hormone, dehydroepiandrosterone (DHEA) and estrogen replacement therapy or placebo, we will determine the effects of an 18-month treatment course on bone mass, circulating markers of bone turnover, and serum levels of a factor, insulin-like growth factor I (IGF-I). We are also studying if these therapies change bone structure to increase skeletal strength compared to placebo, as assessed through cross-sectional geometric analysis of our bone density data by dual-energy x-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
Profound osteopenia is a frequent and often irreversible complication of anorexia nervosa (AN). Adolescents with AN often have a reduced peak bone mass and are at increased risk for early osteoporosis and fractures. These young women have subnormal serum levels of gonadal steroids and the adrenal androgen dehydroepiandrosterone (DHEA) that may be associated with their low bone mineral density (BMD). Low DHEA levels are accompanied by decreased levels of insulin-like growth factor I (IGF-I), estrogen, and testosterone. Previous data from our group indicate that oral DHEA therapy in young women with AN: increases lean body mass, serum levels of bone formation markers and insulin-like growth factor I (IGF-I), and decreases urinary markers of bone resorption. We also found that standard hormonal replacement therapy (HRT) significantly decreased bone resorption markers. Information on the effects of these therapies on bone strength and ultimate fracture risk is lacking.

In this project, we will test the hypothesis that combined therapy with DHEA and estrogen/progestin will enhance bone mass in patients with AN through anabolic and antiosteolytic mechanisms. We will test the hypothesis that 18 months of DHEA + HRT will increase bone mineral density (BMD) and markers of bone formation, while decreasing bone resorption markers in these patients. The proposed study will examine whether restoring normal levels of DHEA and estrogen in these young women will increase bone mass during a critical period for bone accretion. The study will also examine whether DHEA's anabolic effects on bone are mediated through the skeletal IGF-I regulatory system. Using cross-sectional analyses of dual energy x-ray absorptiometry (DXA) data, we will also measure indices of bone structural geometry to determine if mechanical strength is compromised in these young women, and if strength is restored in response to combined anabolic/antiresorptive therapy.

To gain new information on the mechanisms underlying bone loss and fracture risk in young women with AN, our research goals are:

Specific Aim I: Through a randomized controlled trial, to measure the effects of an 18-month course of DHEA + HRT on bone mass, markers of bone turnover, and serum levels of IGF-I compared to placebo. Specific Aim II: To determine whether combined therapy with adrenal and gonadal steroid replacement changes bone structure to increase strength compared to placebo, as assessed through cross-sectional geometric analysis of DXA data.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 - 30 years
* Anorexia nervosa by psychiatric criteria
* Amenorrhea for at least 3 months

Exclusion Criteria:

* Receiving no medications known to affects bone metabolism
* No other chronic medical conditions

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2004-04; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M. Gordon, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vajapeyam S, Ecklund K, Mulkern RV, Feldman HA, O'Donnell JM, DiVasta AD, Rosen CJ, Gordon CM. Magnetic resonance imaging and spectroscopy evidence of efficacy for adrenal and gonadal hormone replacement therapy in anorexia nervosa. Bone. 2018 May;110:335-342. doi: 10.1016/j.bone.2018.02.021. Epub 2018 Feb 26. PMID 29496516
- [Result] Divasta AD, Feldman HA, Brown JN, Giancaterino C, Holick MF, Gordon CM. Bioavailability of vitamin D in malnourished adolescents with anorexia nervosa. J Clin Endocrinol Metab. 2011 Aug;96(8):2575-80. doi: 10.1210/jc.2011-0243. Epub 2011 Jun 1. PMID 21632810
- [Result] Divasta AD, Feldman HA, Gordon CM. Vertebral fracture assessment in adolescents and young women with anorexia nervosa: a case series. J Clin Densitom. 2014 Jan-Mar;17(1):207-11. doi: 10.1016/j.jocd.2013.02.011. Epub 2013 Apr 3. PMID 23562364
- [Result] DiVasta AD, Feldman HA, Beck TJ, LeBoff MS, Gordon CM. Does hormone replacement normalize bone geometry in adolescents with anorexia nervosa? J Bone Miner Res. 2014 Jan;29(1):151-7. doi: 10.1002/jbmr.2005. PMID 23744513
- [Result] DiVasta AD, Mulkern RV, Gordon CM, Ecklund K. MR Imaging in a case of severe anorexia nervosa: the 'flip-flop' effect. Pediatr Radiol. 2015 Apr;45(4):617-20. doi: 10.1007/s00247-014-3145-3. Epub 2014 Aug 17. PMID 25129340
- [Result] Donaldson AA, Feldman HA, O'Donnell JM, Gopalakrishnan G, Gordon CM. Spinal Bone Texture Assessed by Trabecular Bone Score in Adolescent Girls With Anorexia Nervosa. J Clin Endocrinol Metab. 2015 Sep;100(9):3436-42. doi: 10.1210/jc.2015-2002. Epub 2015 Jun 24. PMID 26108094
- [Result] DiVasta AD, Feldman HA, O'Donnell JM, Long J, Leonard MB, Gordon CM. Effect of Exercise and Antidepressants on Skeletal Outcomes in Adolescent Girls With Anorexia Nervosa. J Adolesc Health. 2017 Feb;60(2):229-232. doi: 10.1016/j.jadohealth.2016.10.003. Epub 2016 Dec 6. PMID 27939877
- [Result] DiVasta AD, Feldman HA, O'Donnell JM, Long J, Leonard MB, Gordon CM. Skeletal outcomes by peripheral quantitative computed tomography and dual-energy X-ray absorptiometry in adolescent girls with anorexia nervosa. Osteoporos Int. 2016 Dec;27(12):3549-3558. doi: 10.1007/s00198-016-3685-5. Epub 2016 Jul 8. PMID 27392467
- [Result] Bialo SR, Gordon CM. Underweight, overweight, and pediatric bone fragility: impact and management. Curr Osteoporos Rep. 2014 Sep;12(3):319-28. doi: 10.1007/s11914-014-0226-z. PMID 24986712
- [Result] Ecklund K, Vajapeyam S, Mulkern RV, Feldman HA, O'Donnell JM, DiVasta AD, Gordon CM. Bone marrow fat content in 70 adolescent girls with anorexia nervosa: Magnetic resonance imaging and magnetic resonance spectroscopy assessment. Pediatr Radiol. 2017 Jul;47(8):952-962. doi: 10.1007/s00247-017-3856-3. Epub 2017 Apr 22. PMID 28432403

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Active
Started | 40 | 40
Completed | 30 | 30
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (4) | 24 (6) | 22 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Areal Bone Density by DXA
Time Frame: 18-Months
Measure: Mean (Standard Deviation); unit: g/cm2
Groups:
- Placebo: Sugar Pill
- Active: DHEA+HRT
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 31
g/cm2 | 0.88 (0.10) | 0.89 (0.10)

ADVERSE EVENTS:
Arm/Group | Placebo | Active
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes